CLINICAL TRIAL: NCT01691625
Title: Concurrent Chemoradiation With or Without DC-CIK Immunotherapy in Treating Locally Advanced Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director,Capital Medical University (CMU)Cancer Center,, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-01
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Carcinoma
Keywords: Locally advanced esophageal carcinoma; DC-CIK; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- concurrent chemoradiotherapy plus DC-CIK immunotherapy (Experimental): patients will receive concurrent chemoradiotherapy plur DC-CIK immunotherapy
  Interventions: Other: concurrent chemoradiotherapy plus DC-CIK immunotherapy
- Concurrent chemoradiation only (Active Comparator): patients will receive concurrent chemoradiotherapy only
  Interventions: Other: Concurrent chemoradiation only

INTERVENTIONS:
Other: concurrent chemoradiotherapy plus DC-CIK immunotherapy — Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) or Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-66Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  Chemotherapy: Patients will be concurrently administered with irradiation every 4 weeks with PT regimen (cis-platinum of 20 mg/m2/d, d2-5; PTX(paclitaxel)of 80mg/m2/d, d1,d8) for 4 cycles.The chemotherapy will be concurrently given with irradiation.
  DC-CIK Immunotherapy:Mononuclear cells were collected aseptically with blood cell separator composition apheresis 3 days before concurrent chemoradiation, and cultured DC-CIK cells for 10 days. Cells were infused back to the patients in 3 times between the Chemoradiation intermittent period.
  Arms: concurrent chemoradiotherapy plus DC-CIK immunotherapy
Other: Concurrent chemoradiation only — Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) or Intensity-modulated radiation therapy(IMRT)was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-66Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.
  Chemotherapy: Patients will be concurrently administered with irradiation every 4 weeks with PT regimen (cis-platinum of 20 mg/m2/d, d2-5; PTX(paclitaxel)of 80mg/m2/d, d1,d8) for 4 cycles.The chemotherapy will be concurrently given with irradiation.
  Arms: Concurrent chemoradiation only

SUMMARY:
The purpose of this study is to show if the adoptive cellular therapy with autologous dendritic cells and cytokine-induced killer cells (CIK) combined with concurrent chemoradiation could improve the quality of life of the patients with locally advanced esophageal cancer, compared with concurrent chemoradiation only.

ELIGIBILITY:
Inclusion Criteria:

* cytologically or histologically confirmed locally advanced esophageal carcinoma
* Age: > 18
* Karnofsky performance status ≥ 70
* At least one measurable tumor lesions according to the RECIST criteria.
* Normal functions of heart, lung, liver, kidney and bone marrow
* Blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL
* Informed consent signed

Exclusion Criteria:

* Patients with metastatic disease in the central nervous system (CNS).
* Patients who are pregnant or nursing.
* Patients with poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable
* Patients with contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis
* coexisted morbidities that investigators believed not suitable for chemoradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
the quality of life | initial assessment, months 1, 3, 6 and 12

SECONDARY OUTCOMES:
progression-free survival | 1 year

OTHER OUTCOMES:
Immunological assessment | baseline, months 1, 3, 6 and 12
  Cytokine secretion and T cell populations are assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Cancer Center, Beijing, Beijing Municipality, China